CLINICAL TRIAL: NCT06099613
Title: A Phase I/IIa Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-COVII in Healthy Adult Volunteers
Brief Title: Study to Safety, Tolerability and Immunogenicity of EG-COVII in Healthy Adult
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EyeGene Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: EG-COVID-103
Record Dates: First submitted 2023-10-23; First posted 2023-10-25 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EG-COVII (Experimental)
  Interventions: Biological: EG-COVII

INTERVENTIONS:
Biological: EG-COVII — EG-COVII is a bivalent vaccine to prevent SARS-CoV-2 infection against wild type and Omicron variants

SUMMARY:
This is a Phase I/IIa Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-COVII in Healthy Adult Volunteers

DETAILED DESCRIPTION:
Subjects will undergo a Screening period beginning up to 2 weeks prior to enrollment, the vaccinations will be administered on week 0 and week 3, pre- and post-dose assessment, follow-up visits, and an end of study (EOS) or early termination (ET) visit (as applicable).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure;
* Healthy volunteers aged above 18 years at the time of screening;
* Have had at least authorised primary COVID-19 vaccination(s) regardless of numbers of booster;
* The last authorised COVID-19 vaccination, the participants received, should be more than 16 weeks prior to the first IP vaccination;

Exclusion Criteria:

* Participant with the evidence of COVID-19 infection at screening (Positive for COVID-19 with RT-PCR test with nasal mid-turbinate specimen);
* Participant who has the history of COVID-19 infection within 6 months from the first IP vaccination;
* Close contact with a person infected with COVID-19 within 2 weeks prior to the first IP vaccination;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EG-COVII in healthy adult volunteers | 7 weeks follow up
  Number of participants with adverse events (AEs) Number of participants with abnormal clinical laboratory results (hematology /chemistry /urinalysis) Number of participants with abnormal vital sign Number of participants with abnormal physical examination results

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chang, Dr., Principal Investigator — Nucleus Network Pty Ltd- Melbourne
Locations (1):
- Nucleus Network Pty Ltd- Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No